CLINICAL TRIAL: NCT05618665
Title: The Effect of Education Given to Asthmatic School Children and Their Parents by Taking Health Literacy Into Account on Disease Self-management
Brief Title: The Effect of Asthma Education Given by Taking Health Literacy Into Account
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Esma Guney Kizil, Phd, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-05
Record Dates: First submitted 2022-11-03; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Asthma in Children; Health Literacy; Child Health; Asthma Management; Nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group - Children and parents (Experimental): Asthma education which consisted of asthma disease, its symptoms, diagnosis, treatment, risk factors, use of medication, use of medication apparatus, vaccination treatment, follow-up of the asthmatic child, precautions to be taken in prevention, what to do during an attack, what to do for adaptation to the disease and things to do in school life was prepared and presented in 40 minutes. The booklets about education would be given at the end of the education.
  Interventions: Other: Asthma Education; Other: Delivery of booklets
- Intervention Group - Children (Experimental): Asthma education which consisted of asthma disease, its symptoms, diagnosis, treatment, risk factors, use of medication, use of medication apparatus, vaccination treatment, follow-up of the asthmatic child, precautions to be taken in prevention, what to do during an attack, what to do for adaptation to the disease and things to do in school life was prepared and presented in 40 minutes. The booklets about education would be given at the end of the education.
  Interventions: Other: Asthma Education; Other: Delivery of booklets
- Control group (No Intervention): No intervention was applied to the control group.

INTERVENTIONS:
Other: Asthma Education — Asthma education about asthma disease, its symptoms, diagnosis, treatment, risk factors, use of medication, use of medication apparatus, vaccination treatment, follow-up of the asthmatic child, precautions to be taken in prevention, what to do during an attack, what to do for adaptation to the disease and things to do in school life.
  Arms: Intervention Group - Children; Intervention Group - Children and parents
Other: Delivery of booklets — The booklets, prepared by the researchers, included information about the content of the education.
  Arms: Intervention Group - Children; Intervention Group - Children and parents

SUMMARY:
The aim of this randomized controlled trial was to examine the effect of education given to asthmatic children and their parents by taking health literacy into account on disease self-management.

The study was conducted with 88 children and their parents between October 2018 and July 2019. While education and booklets were given to both children and parents in intervention group 1, only the children were given the education and the booklets in intervention group 2. There was no intervention applied for the control group. Post-test was performed 3 weeks after the education and then follow-ups were carried out in the next three months over the phone.

ELIGIBILITY:
Inclusion Criteria:

* Having asthma children with a physician diagnosis,
* Studying in one of the public primary schools in the district where the study was conducted,
* Using asthma medication,
* Having parents without any reading difficulties.

Exclusion Criteria:

* Being in the 1st grade in their school,
* Not using any medication for asthma,
* Having parents with reading difficulties.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Health Literacy for School-Aged Children - HLSAC | 4 Months
  Health Literacy for School-Aged Children - HLSAC, which was developed by Paakkari et al., is a brief, multidimensional, generic, theory-based, cross-national validated, self-administered instrument to measure the subjective health literacy level of school-aged children. This tool assesses health literacy in five areas among school-aged children: theoretical knowledge (items 1 and 5); practical knowledge (items 4 and 7); critical thinking (items 3 and 9); self-awareness (items 8 and 10), and citizenship (items 2 and 6). The scale items are rated on a four-point Likert-type scale (not at all true = 1, barely true = 2, somewhat true = 3, and absolutely true = 4). A score between 10 and 25 implies low health literacy, between 26 and 35, moderate health literacy, and between 36 and 40, high health literacy.
Health Literacy Scale | 4 Months
  The health literacy levels of the parents were measured with the "Health Literacy Scale". The scale is the short form of the Health Literacy Survey in Europe (HLS-E.U). The scale is a 25-item Health Literacy Index form. The scale consists of 25 items and 4 sub-dimensions: Accessing information (items 1-5), understanding information (items 6-12), valuing/evaluating (items 13-20), and implementing/using (items 21-25). The scale is a 5-point Likert type (1 = I am unable to do / I have no ability / impossible, 2 = I have a lot of difficulties, 3 = I sometimes have difficulties, 4 = I have difficulties, 5 = I have no difficulty). The total score that can be obtained from the scale is between 25 and 125.
Asthma Control Test | 4 Months
  An asthma control test involves questions relating to daytime and nighttime asthma symptoms. This test helps determine if a person is controlling their asthma well. The test helps someone identify how their symptoms interfere with their day-to-day life. If individuals do not have sufficient control over their asthma in the long term, it can increase the risk of asthma attacks and lead to other health issues, such as lung infections, which can cause several symptoms. Five questions involve a 4-week recall of symptoms and how they affect a person's daily functioning. Each answer has a value of 1-5, and at the end of the test, the score for each answer is added to the total score, which may range from 5 to 25. The lower the score, the more a person lacks control of their condition. For example, someone does not have their asthma under control if they score 5 or 6. An individual has better control of their asthma if they score 20 or higher.

CONTACTS AND LOCATIONS:
Overall Officials: Ayla BAYIK TEMEL, Prof., Study Director — Department of Nursing, Ege University
Locations (1):
- Department of Nursing Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No